CLINICAL TRIAL: NCT05136066
Title: Effects of Massage With Diluted Peppermint Oil on Visual Analogue Scoring in Reducing Labor Pain
Brief Title: Effects of Massage With Peppermint Oil on Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Bedir Fındık, Associate Professor Dr, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-MH-RBF-01
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Labor Pain
Keywords: labor pain; mint oil; Visuel anolgue Scoring
MeSH Terms: conditions — Labor Pain | interventions — Massage; peppermint oil

STUDY DESIGN:
Intervention Model Description: Two groups with mint oil control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group massaged with peppermint oil (Experimental): Group of experimental
  Interventions: Other: massage with peppermint oil

INTERVENTIONS:
Other: massage with peppermint oil — Peppermint oil diluted with 1/10 pure olive oil will be applied to the pregnant to reduce labor pain.

SUMMARY:
Birth is a very special experience for a woman and her family. Labor pain is one of the strongest known and defined pains today. In the literature, it has been stated that labor pain is perceived as more severe than chronic pain such as low back pain, cancer pain, phantom pain and postherpetic neuralgia, and acute pain such as fracture or laceration.

When birth pain is not controlled, the vicious cycle of stress, fear and pain can continue and affect the mother and fetus negatively.

In this study, our aim is to determine the effect of applying peppermint oil diluted with pure natural olive oil to the abdomen and waist region by massage in labor pain, reducing the labor pain.

DETAILED DESCRIPTION:
The study is a Prospective Cross-sectional Case Control study. Pregnant women whose mother tongue is Turkish, who are term pregnant and who are in active labor, who are hospitalized in the delivery room of our hospital for delivery, that is, who have a gap of at least 70% 5-6 cm in the examination and who have at least 4-5 severe contractions in 10 minutes, who have a single, vertex-presented fetus will be included in our work. Pregnant women with co-morbidities, chronic diseases, complications related to childbirth, anemic inactive labor, thyroid disease, skin lesions or infections, allergies, multiple pregnancies, use of any medication, and risky pregnancy will be excluded from the study.

For this, 30 pregnant women who were applied peppermint oil and 30 control group pregnant women who were not applied will be included in the study. Following the signed consent form obtained from our patients, visual analog scoring (VAS) will be provided to the patient during the painful period, and then peppermint oil will be applied to the abdomen and lumbar region where he feels the most pain, with 1/10 diluted peppermint oil by hand massage or with the help of a compress moistened with warm water. After the application, visual pain scoring will be applied to pregnant women again.The study is terminated when sufficient data is obtained.

The data will be entered into the computer in the SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* normal pregnant with vertex presentation
* at least 70% 5-6 cm gap in the examination at least 4-5 severe contractions in 10 minutes
* Turkish-speaking

Exclusion Criteria:

* Pregnant women with co-morbidities, chronic diseases
* complications related to childbirth
* inactive labor
* anemic, thyroid disease, skin lesions or infection, allergies, multiple pregnancies
* use of any medication
* risky pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | during labor process, until the labor process is done
  The scale has 0-10 points.As the point increases the pain score increases

CONTACTS AND LOCATIONS:
Overall Officials: Rahime Bedir Findik, Dr, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No